CLINICAL TRIAL: NCT06528080
Title: A Prospective, Single-center, Open-label, Single-arm Clinical Study to Evaluate the Safety and Efficacy of a Single Intravenous Infusion of LY-M001 Injection in Pediatric and Adolescent Patients With Type 1 Gaucher Disease
Brief Title: A Clinical Study for the Treatment of Pediatric and Adolescent Patients With Type 1 Gaucher Disease
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiumin Wang, PhD, Director, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-M001-GD-002
Record Dates: First submitted 2024-06-22; First posted 2024-07-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LY-M001 Backdose (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at backdose.
  Interventions: Genetic: LY-M001
- LY-M001 Dose group 1 (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at dose group 1.
  Interventions: Genetic: LY-M001
- LY-M001 Dose group 2 (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of LY-M001 at dose group 2.
  Interventions: Genetic: LY-M001

INTERVENTIONS:
Genetic: LY-M001 — LY-M001 Injection by Single Intravenous Infusion

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, efficacy, immunogenicity, PD and PK characteristics of LY-M001 injection in children with GD1 aged 6 years ≤ age < 18 years. This study mainly includes the main study stage and the long-term follow-up study stage.

DETAILED DESCRIPTION:
The study planned to enroll 6-9 patients with GD1 for 5 years, with a total of 34 follow-up visits. The main study period was 52 weeks, and the long-term follow-up period was 53 weeks to 5 years after administration.

In this study, three dose groups were preset, and the first subject was enrolled with 1.0× 10^13 vg/kg as the initial dose (the first dose group). After the safety was determined by DLT observation, subsequent subjects were enrolled. Based on safety and efficacy data, it will be decided by SRC discussion to increase to the next dose group.

This is an open clinical study without blindness.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and/or parent, caregiver, or legal representative must be willing and able to provide written informed consent/consent for the study in accordance with applicable regulations and guidelines and comply with all study access and procedures, including the use of any data collection devices that can be used to directly record participant data.
2. Gender is not limited, 6 years old ≤ 18 years old.
3. Patients with double allele mutation of glucocerebrosidase gene (GBA1) and decreased glucocerebrosidase activity were confirmed by laboratory tests and met the clinical manifestations of type I Gaucher disease.
4. Subjects were newly treated or treated patients with type I Gaucher disease; For patients treated with enzyme replacement therapy (ERT) or substrate clearance therapy (SRT) before screening, 5 drug half-lives are required before administration.
5. The subject is willing to participate in all study follow-up and comply with all study procedures and evaluations.
6. The subject must be willing to refrain from donating blood, organs, tissues, or cells at any time after receiving treatment.
7. Pregnant Women (WOCBP) subjects tested negative for pregnancy.

Exclusion Criteria:

1. Positive AAV8 neutralizing antibody (antibody titer > 1:10).
2. Patients with type II or III Gaucher disease (GD2 or GD3), or with suspected Gaucher disease as assessed by the investigator (e.g., subjects with Gaucher disease-related central nervous system manifestations or abnormal electroencephalogram [EEG] examination).
3. Active and progressive bone diseases that are expected to require surgical treatment within the next 6 months.
4. The subjects were judged by the investigator to have idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), thrombocytopenia, anemia, hepatomeglia, splenomeglia, and/or osteoporosis unrelated to GD (bone mineral density z-score ±2).
5. Treatment with an investigational drug in another clinical study within 28 days prior to screening or 5 half-lives, whichever is older.
6. Evidence of a history of clinically significant liver disease or hepatotoxin exposure that meets, but is not limited to, any of the following at the time of screening:

   ① Progressive hepatomegaly larger than 3 times the normal volume;

   ② History of stage 2 or above hepatic fibrosis;

   ③ AST, ALT, or TBIL were 1.5 times higher than the upper limit of normal (ULN);

   ④ Immune hepatitis;

   ⑤ Hepatitis B surface antigen (HBsAg) positive, and hepatitis B virus deoxyribonucleic acid (HBV-DNA) positive (HBV-DNA>10^3 copy number /mL); Or take hepatitis B drugs (such as interferon, lamivudine, adefovir and entecavir); Or hepatitis C virus (HCV) antibody positive.
7. The subject's blood indicators have any of the following:

   ① The hemoglobin value was < 8.0 g/dL;

   ② Platelet count < 40 × 10^9/L.
8. Refractory epilepsy.
9. Human immunodeficiency virus (HIV) antibody positive or treponema syphilis antibody positive.
10. Subjects had significant clinical comorbidities (such as malignant tumors, primary biliary cirrhosis, or autoimmune liver disease) that the investigators believed might affect the study data or confounding the findings.
11. Subjects have received or plan to receive bone marrow transplantation, hematopoietic stem cell transplantation, and/or major organ transplantation, including but not limited to liver transplantation, kidney transplantation, etc.
12. 3 months before screening, subjects received treatment with erythropoietin, whole blood transfusion, or red blood cell transfusion; Or received platelet transfusion 1 month before screening.
13. Allergic to any component of LY-M001 injection.
14. Previous treatment with any type of gene therapy or cell therapy.
15. Use of systemic immunosuppressant or steroid therapy within 3 months prior to administration (other than immunosuppressive therapy prescribed for prophylactic administration).
16. Any condition in which the subject is unable to undergo magnetic resonance imaging (MRI) studies (including hypersensitivity to anesthetics or contrast agents).
17. Have received live attenuated vaccine within 4 months prior to screening or plan to receive live attenuated vaccine during clinical trials.
18. Other situations in which the investigator considers the subject. inappropriate for study participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) and serious adverse events (SAE) within 52 weeks after LY-M001 infusion | Within 52 weeks of infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Incidence rate of dose-limiting toxicity (DLT) events determined by the data safety review committee (SRC) within at least 28 days after LY-M001 infusion | Within 52 weeks of infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.The adverse events defined as dose-limiting toxicity (DLT) have been clearly specified in the protocol.
Liver function levels (including alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin [TBIL], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT]) within 52 weeks after LY-M001 infusion. | Within 52 weeks of infusion
  Incidence rate of liver function-related adverse events evaluated by CTCAE V5.0.

SECONDARY OUTCOMES:
Pharmacodynamics on blood glucocerebrosidase | Within 52 weeks of infusion
  Blood glucocerebrosidase (GCase) protein level and activity level
Pharmacodynamics on Blood glucosesphingosine | Within 52 weeks of infusion
  Blood glucosesphingosine (Lyso-GL1) levels
Effectiveness of symptom improvement on Liver volume | Within 52 weeks of infusion
  Liver volume
Effectiveness of symptom improvement on spleen volume | Within 52 weeks of infusion
  spleen volume
Effectiveness of symptom improvement on Hemoglobin levels | Within 52 weeks of infusion
  Hemoglobin levels
Effectiveness of symptom improvement on platelet counts | Within 52 weeks of infusion
  platelet counts
Effectiveness of symptom improvement on bone mineral density (BMD) after administration | Within 52 weeks of infusion
  Bone mineral density (BMD)
Effectiveness of symptom improvement on bone marrow load (BMB) after administration | Within 52 weeks of infusion
  Bone marrow load (BMB) after administration
Effectiveness of symptom improvement on GD patient Quality of Life scale score | Within 52 weeks of infusion
  GD patient Quality of Life scale score

CONTACTS AND LOCATIONS:
Overall Officials: xiumin wang, PhD, Study Director — Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Shanghai Children's Medical Center, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No